CLINICAL TRIAL: NCT04581265
Title: A Multicenter Phase II Clinical Study of Albumin-bound Paclitaxel (Nab-PTX), Ifosfamide and Cisplatin in the Treatment of Pediatric Advanced, Recurrent or Refractory Extracranial Germ Cell Tumor.
Brief Title: Nab-PTX, Ifosfamide and Cisplatin in the Treatment of Pediatric Extracranial Germ Cell Tumor.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhuo Zhang, Director of department of pediatric cancer,Principal Investigator,Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: nab-PTX-sun
Record Dates: First submitted 2020-09-13; First posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Extracranial Germ Cell Tumor, Pediatric
MeSH Terms: interventions — Albumin-Bound Paclitaxel; Ifosfamide; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nab-PTX, ifosfamide and cisplatin (Experimental): albumin-bound paclitaxel (nab-PTX), ifosfamide and cisplatin in the treatment of pediatric advanced, recurrent or refractory extracranial germ cell tumor.
  Interventions: Drug: albumin-bound paclitaxel (nab-PTX), ifosfamide and cisplatin

INTERVENTIONS:
Drug: albumin-bound paclitaxel (nab-PTX), ifosfamide and cisplatin — Participants received a single dose of albumin-bound paclitaxel (nab-PTX) 270mg/m2/d, administered intravenously (IV) on Day 1; Ifosfamide 1.2g/m2/d administered intravenously (IV) on Day 2-6; Cisplatin 20mg/m2/d administered intravenously (IV) on Day 2-6.

SUMMARY:
The purpose is to evaluate the effectiveness and safety of albumin-bound paclitaxel (nab-PTX), ifosfamide and cisplatin in the treatment of children patients with advanced, recurrent or refractory extracranial germ cell tumor.

DETAILED DESCRIPTION:
Children patients with advanced, recurrent or refractory extracranial germ cell tumor were treated with albumin-bound paclitaxel (nab-PTX), ifosfamide and cisplatin . This is a multi-center and single arm phase II clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 1-18 years old;
2. ECOG PS score: 0-1;
3. Patients was confirmed pathologically with malignant germ cell tumor.
4. Patients with tumor progressed, relapsed or refractory after first-line chemotherapy, and complete or partial remission was not achieved after recent treatment.
5. Have at least one measurable lesion defined by RECIST standard;
6. The estimated survival time was more than 6 months;
7. Patients must fully recover from the acute toxicity of previous anticancer chemotherapy:
8. Bone marrow function met the following criteria:

   1. Absolute neutrophil count (ANC) ≥ 1.0 × 109 / L;
   2. Platelet count ≥ 100.0 × 109 / L (not after platelet transfusion);
9. Liver and kidney function should meet the following criteria:

   1. Bilirubin (the sum of bound and unconjugated) ≤ 1.5 × upper limit of normal value (ULN) (corresponding to age). Patients with confirmed Gilbert's syndrome can be classified according to the researcher;
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN;
   3. Estimated glomerular filtration rate ≥ 70 ml / min / 1.73 m2 or normal serum creatinine (CR);
10. Adequate pulmonary function: no dyspnea at rest, no exercise intolerance, pulse oxygen saturation > 94% (if there are clinical symptoms);
11. Cardiac function:

    1. LVEF ≥ 50% was detected by echocardiography;
    2. There was no history of arrhythmia requiring drug intervention before enrollment;
12. Seizures that can be fully controlled without enzyme-induced anticonvulsants;
13. During the study period, they were able to comply with outpatient treatment, laboratory monitoring and necessary clinical visits;
14. Parents / guardians of child or adolescent subjects have the ability to understand, agree and sign the study informed consent form (ICF) and the applicable child consent form before starting any program related procedures; subject has the ability to express consent (when applicable) with the consent of parents / guardians.

Exclusion Criteria:

Patients with any of the following items will not be enrolled in this study:

1. Patients with recurrent germ cell tumor were treated by surgery alone previously;
2. Patients with immature teratoma (any grade);
3. Patients with sex cord stroma;
4. HBsAg positive patients;
5. Patients with HIV or syphilis infection;
6. Patients who had received organ transplantation before;
7. Uncontrolled active systemic bacterial, viral or fungal infections;

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Estimated)
Dates: Start 2020-11-10 (Estimated); Primary Completion 2023-11-10 (Estimated); Study Completion 2024-05-10 (Estimated)

PRIMARY OUTCOMES:
overall response rate，ORR | From the beginning of observation to the 2 cycles of observation(each cycle is 21 days)
  Percentage of participants who experienced an overall response (overall response rate，ORR) of albumin-binding paclitaxel, ifosfamide, cisplatin regimen in the treatment of advanced, recurrent and refractory children with extracranial germ cell tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhuo Zhang, Principal Investigator — Sun Yat-sen University CancerCenter